CLINICAL TRIAL: NCT04748601
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 4 Study to Evaluate the Efficacy and Safety of Qudexy(R) XR in the Prevention of Migraine in Children 6 to 11 Years of Age
Brief Title: Qudexy XR for the Prevention of Migraine in Children 6 to 11 Years Old
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Upsher-Smith Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P255-501
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Qudexy XR (Experimental)
  Interventions: Drug: Qudexy XR

INTERVENTIONS:
Drug: Qudexy XR — Extended-Release Capsule
  Arms: Qudexy XR
Drug: Placebo — Qudexy XR Matching capsules
  Arms: Placebo

SUMMARY:
A Phase 4 study to evaluate Qudexy XR for the prevention of migraine in children 6 to 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a female or male 6 to 11 years of age, inclusive, at Visit 1 (Screening)
2. Subject weighs at least 17.0 kg and less than 50.0 kg at Visit 1 (Screening) based on 95 percentile weight for the age range.11
3. Subject has at least a 6-month history of headaches consistent with a diagnosis of migraine with or without aura (International Classification of Headache Disorders, 3rd Edition [ICHD 3]).
4. Subject had ≥8 self-reported headache days in the 28 days prior to Screening.
5. Subject has a PedMIDAS score >10, indicating at least mild disruption in daily activities, and <140, indicating extreme disability that may require more comprehensive, multi component therapy.

Exclusion Criteria:

1. Subject has continuous migraines, defined as an unrelenting headache for a 28-day period.
2. Subject is currently receiving treatment or has used Botulinum toxin (Botox®) within 3 months prior to Visit 1 (Screening).
3. Subject is currently receiving migraine prevention medication and has initiated or changed the dose within 28 days of Screening or is unwilling to avoid making a change during the duration of the study.
4. Subject has previously failed an adequate trial of topiramate (at least 3 months duration at a clinically appropriate dose) for prophylaxis of migraine headache due to lack of efficacy or AEs.
5. Subject has previously failed an adequate trial of >3 migraine preventative medications.
6. Subject has a known history of allergic reaction to topiramate or any excipient in Qudexy XR.
7. Subject has a diagnosis or history of disease that may interfere with safety or evaluation of the study drug.
8. Subject is currently using an investigational drug or device or has used such within 30 days prior to Visit 1.
9. Subject has begun menses and any of the following:

   1. Subject has tested positive for pregnancy; OR
   2. Subject is pregnant, planning pregnancy, or lactating; OR
   3. Subject is taking an oral hormonal contraceptive (either combined [estrogen and progestogen containing] or progestogen-only) and is unable or unwilling to switch to an alternative highly effective contraceptive method.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline (last 28 days Run-In Period) in the monthly number of headache days during the 8-week Maintenance Period based on the diary. | 16 Weeks

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Upsher-Smith Clinical Trial Site #5, Birmingham, Alabama
  - Upsher-Smith Clinical Trial Site #15, La Jolla, California
  - Upsher-Smith Clinical Trials Site #3, Aurora, Colorado
  - Upsher-Smith Clinical Trial Site #1, Stamford, Connecticut
  - Upsher-Smith Clinical Trial Site #12, Loxahatchee Groves, Florida
  - Upsher-Smith Clinical Trial Site #8, Orlando, Florida
  - Upsher-Smith Clinical Trial Site #14, Tampa, Florida
  - Upsher-Smith Clinical Trial Site #2, Ann Arbor, Michigan
  - Upsher-Smith Clinical Trial Site #11, Jackson, Mississippi
  - Upsher-Smith Clinical Trial Site #10, Bridgeton, Missouri
  - Upsher-Smith Clinical Trial Site #4, Cincinnati, Ohio
  - Upsher-Smith Clinical Trial Site #6, Portland, Oregon
  - Upsher-Smith Clinical Trials Site #7, Springfield, Oregon
  - Upsher-Smith Clinical Trial Site #13, McAllen, Texas
  - Upsher-Smith Clinical Trial Site #9, Huntington, West Virginia